CLINICAL TRIAL: NCT02890069
Title: Phase Ib, Open-label, Multi-center Study to Characterize the Safety, Tolerability and Pharmacodynamics (PD) of PDR001 in Combination With LCL161, Everolimus (RAD001) or Panobinostat (LBH589)
Brief Title: A Study of PDR001 in Combination With LCL161, Everolimus or Panobinostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X2102
Record Dates: First submitted 2016-05-09; First posted 2016-09-07 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer, Non-small Cell Lung Carcinoma (Adenocarcinoma), Triple Negative Breast Cancer, Renal Cell Carcinoma
Keywords: PDR001; CRC; TNBC; NSCLC; RCC; Immunomodulation; Biomarkers; Bayesian logistic regression model
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma; Triple Negative Breast Neoplasms; Carcinoma, Renal Cell | interventions — spartalizumab; LCL161; Everolimus; Panobinostat; siremadlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- CRC - PDR001 + LCL161 (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: LCL161
- NSCLC - PDR001 + LCL161 (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: LCL161
- TNBC - PDR001 + LCL161 (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: LCL161
- CRC - PDR001+ Everolimus (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: Everolimus
- NSCLC - PDR001+ Everolimus (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: Everolimus
- TNBC - PDR001+ Everolimus (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: Everolimus
- CRC - PDR001 + Panobinostat (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: Panobinostat
- NSCLC - PDR001 + Panobinostat (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: Panobinostat
- TNBC - PDR001 + Panobinostat (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Biological: PDR001; Drug: Panobinostat
- CRC - PDR001 + QBM076 (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Drug: QBM076
- TNBC - PDR001 + QBM076 (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Drug: QBM076
- NSCLC- PDR001 + QBM076 (Experimental): Enrollment to this combination arm is closed to further enrollment.
  Interventions: Drug: QBM076
- CRC - PDR001 + HDM201 (Experimental): Dose escalation completed, expansion arm.
  Interventions: Drug: HDM201
- RCC - PDR001 + HDM201 (Experimental): Dose escalation completed, expansion arm.
  Interventions: Drug: HDM201

INTERVENTIONS:
Biological: PDR001 — anti-PD1 antibody
  Arms: CRC - PDR001 + LCL161; CRC - PDR001 + Panobinostat; CRC - PDR001+ Everolimus; NSCLC - PDR001 + LCL161; NSCLC - PDR001 + Panobinostat; NSCLC - PDR001+ Everolimus; TNBC - PDR001 + LCL161; TNBC - PDR001 + Panobinostat; TNBC - PDR001+ Everolimus
Drug: LCL161
  Arms: CRC - PDR001 + LCL161; NSCLC - PDR001 + LCL161; TNBC - PDR001 + LCL161
Drug: Everolimus
  Other Names: RAD001
  Arms: CRC - PDR001+ Everolimus; NSCLC - PDR001+ Everolimus; TNBC - PDR001+ Everolimus
Drug: Panobinostat
  Other Names: LBH589
  Arms: CRC - PDR001 + Panobinostat; NSCLC - PDR001 + Panobinostat; TNBC - PDR001 + Panobinostat
Drug: QBM076
  Arms: CRC - PDR001 + QBM076; NSCLC- PDR001 + QBM076; TNBC - PDR001 + QBM076
Drug: HDM201
  Arms: CRC - PDR001 + HDM201; RCC - PDR001 + HDM201

SUMMARY:
The purpose of this study was to combine the PDR001 checkpoint inhibitor with several agents with immunomodulatory activity to identify the doses and schedule for combination therapy and to preliminarily assess the safety, tolerability, pharmacological and clinical activity of these combinations.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any procedure
* Patients with advanced/metastatic cancer, with measurable disease as determined by RECIST version 1.1, who have progressed despite standard therapy or are intolerant to SOC, or for whom no standard therapy exists. Patients must fit into one of the following groups:

  • CRC •NSCLC • TNBC• RCC
* ECOG ≤ 2
* Patient must have a site of disease for biopsy, and be a candidate for tumor biopsy according to the institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening, and again during therapy on this study.
* Prior therapy with PD-1/PDL-1 inhibitors is allowed provided any toxicity attributed to prior PD-1- or PD-L1-directed therapy did not lead to discontinuation of therapy.

Exclusion Criteria:

* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy within prior 2 weeks.
* Patients with known hypersensitivity to any of the components of an investigational treatment will be excluded from participation in the corresponding arm but are eligible for participation in other study arm; Patients that have a history of hypersensitivity to rapamycin derivatives will be excluded from participation in the everolimus arm
* History of or current drug-induced interstitial lung disease or pneumonitis grade ≥2
* Out of range lab values as defined in protocol
* Impaired cardiac function or clinically significant cardiac disease
* Active, known or suspected autoimmune disease
* Human Immunodeficiency Virus (HIV), or active Hepatitis C (HCV) virus. Escalation: active Hepatitis B (HBV); Expansion: Patients with Chronic HBV currently on medication will not be excluded.
* Impairment of gastrointestinal (GI) function
* Malignant disease, other than that being treated in this study
* Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity and washout period is 6 weeks; prior immunotherapy - washout is 4 weeks
* Active infection requiring systemic antibiotic therapy.
* Patients requiring chronic treatment with systemic steroid therapy, other than replacement dose steroids or treatment with low, stable dose of steroid (<10 mg/day prednisone or equivalent) for stable CNS metastatic disease.
* Patients receiving systemic treatment with any immunosuppressive medication.
* Major surgery within 2 weeks of the first dose of study treatment
* Radiotherapy within 2 weeks of the first dose of study drug
* Participation in an interventional, investigational study within 2 weeks of the first dose of study treatment.
* Presence of ≥ CTCAE grade 2 toxicity (except alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ CTCAE grade 3) due to prior therapy.
* Use of hematopoietic colony stimulating growth factors </= 3 weeks prior to first dose

Additional exclusion criteria for PDR001/LCL161

* Patients requiring medications metabolized through CYP3A4/5 and have a narrow therapeutic index or medications that are CYP3A4 substrates that cause QT prolongation
* Patients requiring treatment with strong CYP2C8 inhibitors

Additional exclusion criteria for PDR001/Everolimus

* Patients requiring treatment with moderate CYP3A4 inhibitors
* Patients requiring treatment with a strong CYP3A4 inhibitor or inducer

Additional exclusion criteria for PDR001/Panobinostat-

* Patient who received DAC inhibitors
* Patient needing valproic acid during the study or within 5 days prior to first dose
* Patients requiring medications that are sensitive CYP2D6 substrates areCYP2D6 substrates with a narrow therapeutic index or are anti-arrhythmic drugs/drugs with QT-prolongation risks
* Patients requiring a strong inhibitor or inducer of CYP3A4
* Clinically significant, uncontrolled heart disease and/or recent cardiac event within 6 months prior to study
* Unresolved diarrhea ≥ CTCAE grade 2 or a medical condition associated with chronic diarrhea
* Taking medications with QT prolongation risk or interval or inducing Torsade de pointes

Additional exclusion criteria for PDR001/QBM076-

* Patients requiring medications that are strong inducers or strong inhibitors of CYP3A4
* Patients requiring medications with narrow therapeutic index CYP3A4 substrates
* Women using any form of hormonal contraception (oral, injected, implanted, transdermal) will be excluded (unless they are willing to switch to another effective form of contraception under their physician's guidance)

Additional exclusion criteria for PDR001/HDM201-

* Prior treatment with compounds with the same mode of action as proposed for HDM201, i.e. an inhibition of the interaction of TP53 with HDM2, e.g. RG7112 or CGM097
* Patients who require the following treatments moderate to strong CYP3A4 inhibitors; any substrates of CYP3A4/5 with a narrow therapeutic index
* Moderate to strong CYP3A4 inducers
* Patients having out of range values for:

Absolute neutrophil count (ANC) <1500/µL; Platelets < 100 000/µL

Other protocol-defined inclusion exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Phase 1: Incidence of dose limiting toxicities (DLTs) | 5.5 years
  During the first two cycles Cycle = 28 days
Frequency of dose interruptions and reductions | 5.5 years
  Through study completion, an average of 6 months
Frequency and severity of treatment-emergent adverse events (AEs) and serious adverse events (SAEs) | 6 years
  Through study completion, an average of 6 months
Changes between baseline and post-baseline laboratory parameters and vital signs | 6 years
  Through study completion, an average of 6 months
Dose intensities | 6 years
  Through study completion, an average of 6 months

SECONDARY OUTCOMES:
Changes from baseline in ECG parameters in patients recieving PDR001 in combination with Panobinostat | 6 years
  Baseline and end of treatment, an average of 6 months
Best overall response (BOR) | 6 years
  per RECIST v1.1
Time to reach max concentration (Tmax) for PDR001 | 6 years
Presence of anti-PDR001 antibodies | 6 years
Progression free survival (PFS) | 6 years
  per RECIST v1.1
Treatment Free Survival (TFS) | 6 years
Maximum and minimum plasma concentrations of LCL161 (Cmax and Cmin) | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Maximum and minimum Plasma concentrations of everolimus (Cmax and Cmin) | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Maximum and minimum plasma concentrations of panobinostat (Cmax and Cmin) | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Concentration of anti-PDR001 antibodies | 6 years
  Cycle 1 through cycle 6 in treatment period 1 and 2, an average of 6 months
Maximum and minimum serum concentration of PDR001 (Cmax and Cmin) | 6 years
  Cycle 1 through cycle 6 in treatment period 1 and 2, an average of 6 months
Area under the concentration-time curve calculated to the last concentration point (AUClast) for PDR001, as applicable | 6 years
  Cycle 1 through cycle 6 in treatment period 1 and 2, an average of 6 months
Progression free survival (PFS) per irRC | 6 years
Area under the concentration-time curve calculated to the last concentration point (AUClast) for LCL161, as applicable | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Time to reach max concentration (Tmax) for LCL161 | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Time to reach max concentration (Tmax) for Everolimus | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Time to reach max concentration (Tmax) for Panobinostat | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Area under the concentration-time curve calculated to the last concentration point (AUClast) for Everolimus, as applicable | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Area under the concentration-time curve calculated to the last concentration point (AUClast) for Panobinostat, as applicable | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Maximum and minimum Plasma concentrations of QBM076 (Cmax and Cmin) | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Maximum and minimum Plasma concentrations of HDM201 (Cmax and Cmin) | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Time to reach max concentration (Tmax) for QBM076 | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Time to reach max concentration (Tmax) for HDM201 | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Area under the concentration-time curve calculated to the last concentration point (AUClast) for QBM076, as applicable | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months
Area under the concentration-time curve calculated to the last concentration point (AUClast) for HDM201, as applicable | 6 years
  Cycle 1 through cycle 6 in treatment period 1, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- United States (9):
  - UCLA Santa Monica Hematology / Oncology SC, Santa Monica, California
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Regents of the University of Michigan, Ann Arbor, Michigan
  - Washington University Medical School SC, St Louis, Missouri
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - UT Health San Antonio Mays Cancer Center, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Germany (3):
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
- Netherlands (4):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Utrecht
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan
- United Kingdom (3):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18008